CLINICAL TRIAL: NCT00483314
Title: Homocystinuria: Treatment With N-Acetylcysteine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: March of Dimes (Other)
Responsible Party: Brian M. Gilfix, Principal Investigator, McGill University Health Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6-FY06-317
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 2 g p.o. BID x 60 days
  Other Names: NAC

SUMMARY:
The purpose of this study is determine if oral N-acetylcysteine is effective in lowering homocysteine in individuals with homocystinuria.

DETAILED DESCRIPTION:
Homocystinuria (MIM 236200) due to CBS deficiency is the most common inborn error of sulfur amino acid metabolism with severe clinical manifestations. We propose:

1. An open-label pilot study of N-acetylcysteine (NAC) to lower plasma homocysteine levels in those that have not responded to conventional treatment which includes betaine (Cystadane®, Orphan Medical Inc.), which while lowering Hcy levels does not normalize it, and is very expensive. There are no known contraindications to NAC used for nutritional supplementation and it is relatively inexpensive.

   Oral NAC has reduced total plasma homocysteine in healthy subjects in a dose-dependent fashion.
2. Measurement of flow-mediated vasodilation of the brachial artery (endothelial function) in response to NAC treatment. Endothelial dysfunction is a precursor of atherogenesis.
3. Sequencing the CBS gene in these individuals in order to identify novel mutations causing homocystinuria and identify polymorphisms in other genes that may affect response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Homocystinuria (lens dislocation and hyperhomocysteinemia)
* Age ≥ 18 (the age of majority in Canada)

Exclusion Criteria:

* Nursing mothers or pregnant women
* Chronic liver disease
* Taking nitrates
* Cystine stone formers
* History of active peptic ulcer disease
* Subjects receiving carbamazepine and metoclopramide
* Use of other products containing cysteine or N-acetylcysteine (e.g. nebulized NAC, cysteine supplements, methionine restriction)
* Hypersensitivity to any ingredient in the study product
* Clinically significant, abnormal laboratory test on screening (Visit 2)

Other Criteria:

* Women of child-bearing capacity must be using an acceptable method of birth control and have a negative pregnancy test before being enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Lowering plasma total homocysteine | 3 months

SECONDARY OUTCOMES:
Change in flow-mediated dilatation of brachial artery | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian M GILFIX, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - MUHC-Royal Victoria Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- See also: funding agency — http://www.marchofdimes.org